CLINICAL TRIAL: NCT02911922
Title: Randomized Trial of Image -Guided Stereotactic Radiation Therapy (IG-SRT) in Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patient accruals.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1604017139
Record Dates: First submitted 2016-09-19; First posted 2016-09-22 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endorectal balloon - Radiation therapy (Experimental): Group 1 : Endorectal balloon (ERB): Immobilization device manually placed into the rectum prior to radiation treatment planning CT and daily treatment delivery, to immobilize the prostate and reduce prostate motion.
  Patients on each arm will receive 5 fractions of radiation, 7.25Gy per fraction, delivered 2-3 times a week (every other day excluding weekends), to total dose of 36.25 Gy. The total duration of treatment will be no shorter than 10 days.
  Interventions: Device: Endorectal Balloon; Radiation: Radiation therapy
- Rectal spacer - Radiation therapy (Experimental): Group 2 : Rectal spacer (RS): Biodegradable gel that is transperineally injected between the rectum and prostate under transrectal ultrasound guidance, to increase physical distance and thereby reduce radiation dose to the anterior rectal wall. The spacer begins to biodegrade in 2-3 months, and is fully absorbed within 6 months.
  Patients on each arm will receive 5 fractions of radiation, 7.25Gy per fraction, delivered 2-3 times a week (every other day excluding weekends), to total dose of 36.25 Gy. The total duration of treatment will be no shorter than 10 days.
  Interventions: Device: Rectal Spacer; Radiation: Radiation therapy

INTERVENTIONS:
Device: Endorectal Balloon — Endorectal balloon (ERB): Immobilization device manually placed into the rectum prior to radiation treatment planning CT and daily treatment delivery, to immobilize the prostate and reduce prostate motion.
  Patients on each arm will receive 5 fractions of radiation, 7.25Gy per fraction, delivered 2-3 times a week (every other day excluding weekends), to total dose of 36.25 Gy. The total duration of treatment will be no shorter than 10 days.
  Arms: Endorectal balloon - Radiation therapy
Device: Rectal Spacer — Rectal spacer (RS): Biodegradable gel that is transperineally injected between the rectum and prostate under transrectal ultrasound guidance, to increase physical distance and thereby reduce radiation dose to the anterior rectal wall. The spacer begins to biodegrade in 2-3 months, and is fully absorbed within 6 months.
  Patients on each arm will receive 5 fractions of radiation, 7.25Gy per fraction, delivered 2-3 times a week (every other day excluding weekends), to total dose of 36.25 Gy. The total duration of treatment will be no shorter than 10 days.
  Arms: Rectal spacer - Radiation therapy
Radiation: Radiation therapy — Patients on each arm will receive 5 fractions of radiation, 7.25Gy per fraction, delivered 2-3 times a week (every other day excluding weekends), to total dose of 36.25 Gy. The total duration of treatment will be no shorter than 10 days.

SUMMARY:
Patients with low-risk or favorable intermediate-risk prostate cancer as defined by 1.2016 NCCN criteria will be eligible to participate on this study.

DETAILED DESCRIPTION:
This is a randomized, two arm study for patients with low-risk or favorable intermediate-risk prostate cancer as defined by 1.2016 NCCN criteria.

Patients will be randomized to either rectal spacer placement or endorectal balloon placement, daily prior to each radiation treatment.

1. Endorectal balloon (ERB): Immobilization device manually placed into the rectum prior to radiation treatment planning CT and daily treatment delivery, to immobilize the prostate and reduce prostate motion.
2. Rectal spacer (RS): Biodegradable gel that is transperineally injected between the rectum and prostate under transrectal ultrasound guidance, to increase physical distance and thereby reduce radiation dose to the anterior rectal wall. The spacer begins to biodegrade in 2-3 months, and is fully absorbed within 6 months.

This study plans to enroll a total of 40 patients with an accrual period of 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven diagnosis of prostate adenocarcinoma, diagnosed within 1 year of randomization
* Either NCCN-defined low-risk disease (T1c-T2a, Gleason score 3+3=6, PSA <10), intermediate-risk disease (Gleason score 3+4=7, 4+3=7, T2b-c and/or PSA 10-20; ) or high-risk disease due to Gleason score 8-10 and/or PSA >20 ng/ml, but not due to T3-T4 disease on physical exam.

Exclusion Criteria:

* History of prior pelvic radiation (external beam or brachytherapy)
* Prior or concurrent lymphomatous/hematogenous malignancy, or history of prior/concurrent invasive malignancy during the past 5 years
* Very high risk prostate cancer (T3b-T4 on clinical exam, Primary Gleason pattern 5, or >4 cores with Gleason score 8-10)
* History of prior chemotherapy for prostate cancer
* History of irritable bowel disease
* Evidence of lymph node involvement
* AUA score >15
* Prostate size > 90 cc

Ages: 19 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-09; Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Kang, M.D., Principal Investigator — Weill Cornell Medicine - New York Presbyterian Hospital; Silvia Formenti, M.D., Principal Investigator — Weill Cornell Medicine - New York Presbyterian Hospital
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One patient was enrolled on this study overall.
Groups:
- Endorectal Balloon - Radiation Therapy: Group 1 : Endorectal balloon (ERB): Immobilization device manually placed into the rectum prior to radiation treatment planning CT and daily treatment delivery, to immobilize the prostate and reduce prostate motion.Patients on each arm will receive 5 fractions of radiation, 7.25Gy per fraction, delivered 2-3 times a week (every other day excluding weekends), to total dose of 36.25 Gy. The total duration of treatment will be no shorter than 10 days.
  Endorectal Balloon: Endorectal balloon (ERB): Immobilization device manually placed into the rectum prior to radiation treatment planning CT and daily treatment delivery, to immobilize the prostate and reduce prostate motion.Patients on each arm will receive 5 fractions of radiation, 7.25Gy per fraction, delivered 2-3 times a week (every other day excluding weekends), to total dose of 36.25 Gy. The total duration of treatment will be no shorter than 10 days.
- Rectal Spacer - Radiation Therapy: Group 2 : Rectal spacer (RS): Biodegradable gel that is transperineally injected between the rectum and prostate under transrectal ultrasound guidance, to increase physical distance and thereby reduce radiation dose to the anterior rectal wall. The spacer begins to biodegrade in 2-3 months, and is fully absorbed within 6 months.
  Rectal Spacer: Rectal spacer (RS): Biodegradable gel that is transperineally injected between the rectum and prostate under transrectal ultrasound guidance, to increase physical distance and thereby reduce radiation dose to the anterior rectal wall. The spacer begins to biodegrade in 2-3 months, and is fully absorbed within 6 months.
Period: Overall Study
Arm/Group | Endorectal Balloon - Radiation Therapy | Rectal Spacer - Radiation Therapy
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study accrued only one patient . 0(zero) subjects were analyzed in the rectal spacer arm due to lack of accrual.
Groups:
- Endorectal Balloon - Radiation Therapy: Group 1 : Endorectal balloon (ERB): Immobilization device manually placed into the rectum prior to radiation treatment planning CT and daily treatment delivery, to immobilize the prostate and reduce prostate motion.Patients on each arm will receive 5 fractions of radiation, 7.25Gy per fraction, delivered 2-3 times a week (every other day excluding weekends), to total dose of 36.25 Gy. The total duration of treatment will be no shorter than 10 days.
  Endorectal Balloon: Endorectal balloon (ERB): Immobilization device manually placed into the rectum prior to radiation treatment planning CT and daily treatment delivery, to immobilize the prostate and reduce prostate motion.
  Patients on each arm will receive 5 fractions of radiation, 7.25Gy per fraction, delivered 2-3 times a week (every other day excluding weekends), to total dose of 36.25 Gy. The total duration of treatment will be no shorter than 10 days.
- Rectal Spacer - Radiation Therapy: Group 2 : Rectal spacer (RS): Biodegradable gel that is transperineally injected between the rectum and prostate under transrectal ultrasound guidance, to increase physical distance and thereby reduce radiation dose to the anterior rectal wall. The spacer begins to biodegrade in 2-3 months, and is fully absorbed within 6 months.
  Patients on each arm will receive 5 fractions of radiation, 7.25Gy per fraction, delivered 2-3 times a week (every other day excluding weekends), to total dose of 36.25 Gy. The total duration of treatment will be no shorter than 10 days.
  Rectal Spacer: Rectal spacer (RS): Biodegradable gel that is transperineally injected between the rectum and prostate under transrectal ultrasound guidance, to increase physical distance and thereby reduce radiation dose to the anterior rectal wall. The spacer begins to biodegrade in 2-3 months, and is fully absorbed within 6 months.
- Total: Total of all reporting groups
Arm/Group | Endorectal Balloon - Radiation Therapy | Rectal Spacer - Radiation Therapy | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 70 [70 to 70] |  | 70 [70 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1
Health Related Quality of Life Based on Expanded Prostate Cancer Index Composite Question [Number; unit: units on a scale] — Measure the effect of treatment on patients using Health related Quality of Life based on Expanded Prostate Cancer Index Composite Question. For EPIC GU, EPIC GI and Sexual Health higher (range 0-100) scores represent Good quality of life. For AUA scores ( range 0-35), Lower scores represent less urinary symptoms.
  units on a scale
    EPIC GU | 93.8 |  | 93.8
    EPIC GI | 100 |  | 95.8
    EPIC Sexual health | 100 |  | 100
    AUA scores | 6 |  | 6
Comparing Neutrophil:Lymphocyte ratio [Number; unit: Ratio] | 2.23 |  | 2.23

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Patient-reported Acute Toxicity Based on the Common Terminology Criteria for Adverse Events (CTCAE) Version 4
Description: To compare acute toxicity (as defined by CTCAE v4.0) and to compare Rectal dose (V35, max rectal dose). Acute radiation toxicities are side effects that occur on treatment or in the immediate post treatment period (within 90 days from the start of radiation treatment).
Time Frame: Baseline to 1 year
Population: Data was not collected for the Rectal Spacer - Radiation Therapy arm because the trial was terminated due to lack of accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Endorectal Balloon - Radiation Therapy | Rectal Spacer - Radiation Therapy
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

2. Secondary Outcome: Measure the Effect of Treatment on Patients' Using Health Related Quality of Life Based on Expanded Prostate Cancer Index Composite Questionnaire
Description: To compare health-related quality of life (HRQOL) measured using the Expanded Prostate Cancer Index Composite (EPIC) instrument for bowel, urinary and sexual domains. scores are transformed linearly to a 0-100 scale (see following page: EPIC scoring), with higher scores representing better HRQOL. American Urological Association (AUA) scores ranges from 0-30 scores where, score greater than 15 indicate high degree of urinary symptoms and scores less than 15 indicate low degree of urinary symptoms.
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: units on a scale
Arm/Group | Endorectal Balloon - Radiation Therapy | Rectal Spacer - Radiation Therapy
Number analyzed (Participants) | 1 | 0
units on a scale
  EPIC GU (post treatment) | 100 |
  EPIC GI (post treatment) | 95.8 |
  EPIC Sexual health | NA — Patient decline to answer |
  AUA scores | 2 |

3. Secondary Outcome: Number of Participants With Recurrence-free Survival
Description: 1 year
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Endorectal Balloon - Radiation Therapy | Rectal Spacer - Radiation Therapy
Number analyzed (Participants) | 1 | 0
Participants
  Baseline visit | 1 |
  1 month post Radiation visit | 1 |
  6 month post Radiation visit | 1 |
  1 year post Radiation visit | 1 |

4. Secondary Outcome: Comparing Several Parameters That Are Involved in Treatment Planning in Patients Randomized to Two Radiation Therapy Modalities.
Description: To compare the dose distribution of the 2 techniques, specifically:
  1. coverage of the PTV
  2. DVH of organs at risk (OAR)
  3. prostate motion and shifts required during treatment
Time Frame: 5 years
Population: Data could not be analyzed for the secondary outcome measure as we needed more than one patient to compare two radiation techniques. The trial was terminated due to lack of accrual.
Arm/Group | Endorectal Balloon - Radiation Therapy | Rectal Spacer - Radiation Therapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Incidence of Patient-reported Toxicity (Late Toxicity) Based on the Common Terminology Criteria for Adverse Events (CTCAE) Version 4
Description: To compare late toxicity (as defined by CTCAE v4.0). Late toxicities are toxicities that occur greater than 3 months after radiation therapy completion.
Time Frame: post RT to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Endorectal Balloon - Radiation Therapy | Rectal Spacer - Radiation Therapy
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

6. Other Pre Specified Outcome: Measuring Number of Participants Changes in the Microbiome That is Associated With Normal Tissue Toxicities Resulting From Radiation From Baseline to End of Treatment
Description: To explore microbiome changes associated with normal tissue toxicities resulting from radiation
Time Frame: baseline, post radiation follow up
Population: Data was not collected for both Endorectal balloon arm and the Rectal Spacer - Radiation Therapy arm.
Arm/Group | Endorectal Balloon - Radiation Therapy | Rectal Spacer - Radiation Therapy
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Comparing Neutrophile:Lymphocyte Ratio (NLR) at Different Time Points to Assess Impact of SBRT in All the Participants
Description: Comparing NLR ratio at different timepoints to assess the impact of radiation therapy on patients. A neutrophil:lymphocyte ratio (NLR) > 4 at time radiotherapy predicts for significantly worse prognosis, when compared to NLR < 4.
Time Frame: 1 month, 6 months, 1 year
Population: as for outcome 1
Measure: Number; unit: ratio
Arm/Group | Endorectal Balloon - Radiation Therapy | Rectal Spacer - Radiation Therapy
Number analyzed (Participants) | 1 | 0
ratio
  1 month post radiation | 2.4 |
  6 month post radiation | 1.9 |
  1 year post (not collected) | NA — NLR was not collected at this time point. |

ADVERSE EVENTS:
Time Frame: The adverse events were collected over a time period of 1 year.
Description: The adverse events were collected based on the CTCAEv4.03. 0 subjects at risk in the rectal spacer - radiation therapy arm because the trial was closed due to lack of accrual.
Arm/Group | Endorectal Balloon - Radiation Therapy | Rectal Spacer - Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT02911922/Prot_SAP_000.pdf